CLINICAL TRIAL: NCT01743742
Title: The First-day High Dose Vitamin E and Vitamin C in Hypoxic Ischemic Encephalopathy (Following Birth Asphyxia) in Newborns
Brief Title: First-day High Dose Vitamin C, E in Severe Birth Asphyxia
Acronym: CEBA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Takhtasinhji General Hospital (Other Government)
Responsible Party: Principal Investigator, Jayendra R. Gohil, MD, PROF., Professor of Pediatrics, Sir Takhtasinhji General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Antioxidants in Birth Asphyxia
Record Dates: First submitted 2012-11-29; First posted 2012-12-06 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Birth Asphyxia
Keywords: Oral vitamin C and Oral vitamin E
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Vitamin E; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral vitamin E, vitamin C (Experimental): Single dose of vitamin E drops 200 IU within 6 hours of birth and vitamin C tablet 250 mg in pulverised form (2 doses at 24 hr interval) via infant feeding tube
  Interventions: Drug: Vitamin E, Vitamin C

INTERVENTIONS:
Drug: Vitamin E, Vitamin C
  Other Names: Evion® drops; Tablet Limcee®

SUMMARY:
To study the role of first-day high dose oral vitamin C and first-day single high dose oral vitamin E in hypoxic-ischemic encephalopathy in newborns, in the reduction of morbidity and adverse neurodevelopmental sequelae.

DETAILED DESCRIPTION:
Design: A prospective, randomized controlled trial over 5 months. Patients: Newborns admitted within 6 hours after birth with gestation >32 weeks, Apgar score of <6 at 5 minutes, features suggestive of neonatal encephalopathy.

Intervention: After randomization, Group A newborns received oral vitamin C 250 mg once a day within a 24-hour interval along with a single dose of vitamin E 200 IU. Group B newborns received no intervention.

Outcome measures: Severity and progression of birth asphyxia, duration of hospitalization and mechanical ventilation, mortality, and neurodevelopmental outcome.

ELIGIBILITY:
Inclusion Criteria

1. Apgar score of <6 at 5 minutes
2. Clinical features suggestive of neonatal encephalopathy (coma, seizures or hypotonia)

Exclusion Criteria

1. Newborn hospitalized in neonatal intensive care unit (NICU) after 6 hours of birth
2. Gestational age <32 weeks.
3. Lethal congenital anomaly

Ages: 1 Minute to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To assess the role of first day high-dose vitamin E and vitamin C in reduction of adverse neurodevelopmental sequel in newborns with birth asphyxia. | 6 months
  Vitamin C and E were initiated orally within 6 hours of birth.

SECONDARY OUTCOMES:
Mortality and morbidity in newborns with birth asphyxia administered vitamin E and vitamin C. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 15 DAYS.
  Deaths and Sequel were measured.

OTHER OUTCOMES:
Role of single high dose vitamin E and vitamin C in progression or resolution of Hypoxic ischemic encephalopathy. | at 12 hours
  progression of birth asphyxia in terms of HIE Sarnat grading.
Role of single high dose vitamin E and vitamin C in progression or resolution of Hypoxic-ischemic encephalopathy. | 15 days
  Grading of HIE and discharge or death and sequel at followup.

CONTACTS AND LOCATIONS:
Overall Officials: Jayendra R Gohil, MD, Principal Investigator — Professor Pediatrics, Govt Medical College, Bhavnagar, Gujarat, India
Locations (1):
- NICU, Sir T Hospital, Bhavnagar, Bhavnagar, Gujarat, India

REFERENCES:
- [Result] Darlow BA, Buss H, McGill F, Fletcher L, Graham P, Winterbourn CC. Vitamin C supplementation in very preterm infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2005 Mar;90(2):F117-22. doi: 10.1136/adc.2004.056440. PMID 15724034